CLINICAL TRIAL: NCT03482882
Title: An Open-label, 8-Week Study of Safety and Efficacy of Pimavanserin Treatment in Adults With Parkinson's Disease and Depression
Brief Title: Safety and Efficacy of Pimavanserin in Adults With Parkinson's Disease and Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-048
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Treatment of Depression in Adults With Parkinson's Disease (PD)
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Drug - pimavanserin (Experimental)
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg total daily dose, tablets, once daily by mouth (provided as two 17 mg NUPLAZID® tablets)

SUMMARY:
The purpose of this study is to assess the efficacy of pimavanserin for the treatment of depression in adults with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Can understand and provide signed informed consent, request for medical records and/or subject privacy form if applicable according to local regulations
2. Has a clinical diagnosis of idiopathic Parkinson's disease with a minimum duration of 1 year, defined as the presence of at least three of the following cardinal features, in the absence of alternative explanations or atypical features:

   1. rest tremor
   2. rigidity
   3. bradykinesia and/or akinesia
   4. postural and gait abnormalities
3. Meets clinical criteria for depression with Parkinson's disease as listed in the NINDS/NIMH Guidelines
4. If currently taking an anti-depressant, is being treated with only one SSRI or SNRI antidepressant at a dose within the US FDA-approved dose range. Subjects who are currently taking a second antidepressant or antidepressant augmentation agent at a sub-therapeutic dose or for an inadequate duration at Screening, and can be discontinued from this agent before the Baseline visit (in the opinion of the Investigator), may be eligible for the study.
5. Is on a stable dose of anti-Parkinson's medication for 1 month prior to Screening
6. If the subject is female, she must be of non-childbearing potential or agree to use two methods of clinically acceptable contraception

Exclusion Criteria:

1. Use of an antipsychotic within 3 weeks or 5 half-lives of Baseline (whichever is longer)
2. Had a myocardial infarction within the 6 months prior to Screening
3. Has a known personal or family history or symptoms of long QT syndrome
4. Evidence of severe or medically significant hepatic or renal impairment on laboratory tests as assessed by the Investigator or Medical Monitor
5. Has a history of PD psychosis, schizophrenia, or other psychotic disorder, or bipolar I or II disorder.
6. Actively suicidal at Visit 1 (Screening) or Visit 2 (Baseline)
7. Is pregnant or breastfeeding
8. Has previously been treated with pimavanserin or is currently taking pimavanserin
9. Has a sensitivity to pimavanserin or its excipients
10. Is judged by the Investigator or the Medical Monitor to be inappropriate for the study

Additional inclusion/exclusion criteria apply. Subjects will be evaluated at screening to ensure that all criteria for study participation are met.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - ATP Clinical Research, Inc., Costa Mesa, California
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - SC3 Research-Reseda, Pasadena, California
  - The Neurology Group, Pomona, California
  - SC3 Research-Reseda, Reseda, California
  - CNS Network, Torrance, California
  - Associated Neurologists, P.C., Danbury, Connecticut
  - Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Tallahassee Neurological Clinic, P.A., Tallahassee, Florida
  - SRI Biosciences, Clinical Trials and Strategic Development Services, Plymouth, Michigan
  - Washington University School of medicine, St Louis, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - David L. Kreitzman, MD, PC, Commack, New York
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Neurology/Neurophysiology, Johnstown, Pennsylvania
  - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeKarske D, Alva G, Aldred JL, Coate B, Cantillon M, Jacobi L, Nunez R, Norton JC, Abler V. An Open-Label, 8-Week Study of Safety and Efficacy of Pimavanserin Treatment in Adults with Parkinson's Disease and Depression. J Parkinsons Dis. 2020;10(4):1751-1761. doi: 10.3233/JPD-202058. PMID 32804101

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimavanserin: Pimavanserin 34 mg, taken as 2 tablets of pimavanserin 17 mg as a single dose once daily
Period: Overall Study
Arm/Group | Pimavanserin
Started | 47
Completed | 40
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 2
Not completed — Not further specified | 1

BASELINE CHARACTERISTICS:
Population: Patients treated with study drug
Groups:
- Pimavanserin Safety Analysis Set: The Safety Analysis Set (SAS) includes all subjects (47 participants) who received at least one dose of study drug (34mg pimavanserin taken as two 17mg tablets, once daily by mouth)
Arm/Group | Pimavanserin Safety Analysis Set
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 43
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 47
Duration of Parkinson's Disease (PD) [Mean (Standard Deviation); unit: years] | 7.8 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in HAMD-17 (Hamilton Depression Scale -17 Items) Total Score
Description: The HAMD-17 is a multiple-item questionnaire to assess the severity of depression, including items of mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Each of the 17 items is scored on a 3- or 5-point scale (depending on the item). The minimum total score is 0; the maximum total score is 52. A higher total score signifies more severe depression.
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17. The Full Analysis Set had 45 participants at baseline. The Full Analysis Set at Week 8 had 39 participants.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Pimavanserin Full Analysis Set: The Full Analysis Set (FAS) includes all subjects (45 participants) who received at least one dose of study drug (34mg pimavanserin taken as two 17mg tablets, once daily by mouth) and who have both a baseline value and post-baseline value for the Hamilton Depression Scales (17 items; HAMD-17)
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline HAMD-17 total score | 19.2 (0.46)
  Week 8 HAMD-17 total score: number analyzed (Participants) | 39
  Week 8 HAMD-17 total score | 8.1 (0.77)
Statistical Analysis 1: Comparison: Pimavanserin Full Analysis Set; Test type: Other; p < 0.0001, Mixed-effect model repeated measures; LSM = -10.8, 95% CI 2-sided [-12.0 to -9.5], Standard Error of Mean 0.63

2. Secondary Outcome: Change From Baseline (CFB) in HAMD-17 Total Score at Weeks 2, 4, and 6
Description: as for outcome 1
Time Frame: 2, 4, and 6 weeks from baseline
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline HAMD-17 total score | 19.2 (0.46)
  Week 2 HAMD-17 total score CFB: number analyzed (Participants) | 43
  Week 2 HAMD-17 total score CFB | -7.5 (0.89)
  Week 4 HAMD-17 total score CFB: number analyzed (Participants) | 39
  Week 4 HAMD-17 total score CFB | -9.7 (0.69)
  Week 6 HAMD-17 total score CFB: number analyzed (Participants) | 39
  Week 6 HAMD-17 total score CFB | -9.6 (0.69)

3. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I)
Description: The CGI-I is a clinician-rated 7-point scale to rate the improvement in the patient's depression at the time of assessment relative baseline. The CGI-I ranges from 1 (very much improved) to 7 (very much worse)
Time Frame: At Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 39
score on a scale | 2.0 (0.16)

4. Secondary Outcome: Change From Baseline (CFB) in Clinical Global Impression-Severity (CGI-S)
Description: The CGI-S is a clinician-rated 7-point scale to rate the severity of the patient's depression at the time of assessment. The CGI-S ranges from 1 (normal) to 7 (patient is among the most severely ill).
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline CGI-S | 4.1 (0.08)
  8 Week CGI-S CFB: number analyzed (Participants) | 39
  8 Week CGI-S CFB | -1.8 (0.17)

5. Secondary Outcome: Change From Baseline (CFB) in Scale of Outcomes in PD-Sleep Scale (SCOPA) Nighttime Sleep (NS)Score
Description: The SCOPA-NS subscale addresses problems in nighttime sleep and consists of 5 items (sleep initiation, sleep fragmentation, sleep efficiency, sleep duration, early wakening). Each item has 4 response options (ranging from 0=not at all to 3=a lot). The SCOPA-NS score ranges from 0 to 15, with a higher score indicating more severe nighttime sleep problems.
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline SCOPA-NS | 6.1 (0.51)
  Week 8 SCOPA-NS CFB: number analyzed (Participants) | 39
  Week 8 SCOPA-NS CFB | -2.1 (0.57)

6. Secondary Outcome: Change From Baseline (CFB) in SCOPA Daytime Sleepiness (DS) Score
Description: The SCOPA-DS subscale addresses problems in daytime sleepiness and consists of 6 items (falling asleep unexpectedly, falling asleep peacefully, falling asleep watching TV/reading, falling asleep while talking to someone, having difficulty staying awake, whether falling asleep in the daytime is considered a Problem). Each item has 4 response options (from 0=never to 3=often). The SCOPA-DS subscale score ranges from 0 to 18, with a higher score indicating more severe DS problems.
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline SCOPA-DS | 5.2 (0.56)
  8 Week SCOPA-DS CFB: number analyzed (Participants) | 39
  8 Week SCOPA-DS CFB | -2.2 (0.50)

7. Secondary Outcome: The Number (or Percentage) of Responders
Description: The HAMD-17 is a multiple-item questionnaire to assess the severity of depression, including items of mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Each of the 17 items is scored on a 3- or 5-point scale (depending on the item). The minimum total score is 0; the maximum total score is 52. A higher total score signifies more severe Depression.
  Response was defined as ≥50% reduction from baseline in HAMD-17 total score. Patients without Week-8 score were counted as nonresponders.
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
Participants | 27

8. Secondary Outcome: Change From Baseline in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Description: The EQ-5D-5L is a standardized measure of health status. The questionnaire consists of 2 components: the EQ-5D-5L descriptive system and the EQ-5D-5L Visual Analogue scale (EQ-5D-5L VAS). The descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels (from 1=no problem to 5=extreme Problems). The digits for the 5 dimensions are combined into a 5-digit code that describes the patient's health state, which is then converted into a single summary index value. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
  The EQ-5D-5L VAS records the patient's health on a vertical visual analogue scale, ranging from 100 (=the best health you can imagine) to 0 (=the worst health you can imagine).
Time Frame: From baseline to Week 8
Population: Patients treated with study drug and with at least one post-baseline assessment of the HAMD-17
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin Full Analysis Set
Number analyzed (Participants) | 45
score on a scale
  Baseline EQ-5D-5L index score | 0.6750 (0.02551)
  8 Week EQ-5D-5L index score CFB: number analyzed (Participants) | 38
  8 Week EQ-5D-5L index score CFB | 0.0712 (0.02629)
  Baseline EQ-5D-5L VAS | 63.9 (2.43)
  8 Week EQ-5D-5L VAS CFB: number analyzed (Participants) | 38
  8 Week EQ-5D-5L VAS CFB | 6.7 (2.61)

ADVERSE EVENTS:
Time Frame: From the time of informed consent through a safety follow-up visit at Week 10
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47
Other Adverse Events (participants affected / at risk) | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=47)
Colitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=47)
Nausea (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypertonia (Nervous system disorders) | 1 (1)
Mental impairment (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 1 (1)
Illusion (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Rapid eye movement sleep behaviour disorder (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03482882/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/82/NCT03482882/SAP_001.pdf